CLINICAL TRIAL: NCT04344379
Title: Randomized Multicenter Study Evaluating the Efficacy of Azithromycin and Hydroxychloroquine in the Prevention of SARS-CoV-2 Infection in the Hospital Population Exposed to Virus
Brief Title: Prevention of SARS-CoV-2 in Hospital Workers s Exposed to the Virus
Acronym: PREP-COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APHP200386; 2020-001273-73 (EudraCT Number)
Record Dates: First submitted 2020-03-27; First posted 2020-04-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2; hydroxychloroquine; azithromycin; caregivers
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm Title : hydroxychloroquine (Active Comparator)
- Placebo of hydroxychloroquine (Placebo Comparator)
  Interventions: Drug: hydroxychloroquine placebo
- azythromycin (Active Comparator)
  Interventions: Drug: azithromycin

INTERVENTIONS:
Drug: hydroxychloroquine — 200 mg BID per day
Drug: azithromycin — 250 mg per day
  Arms: azythromycin
Drug: hydroxychloroquine placebo — 200 mg BID per day
  Arms: Placebo of hydroxychloroquine

SUMMARY:
The Investigators propose to set up a preventive trial of infection in hospital workers at risk of coronavirus infection by comparing the rate of SARS-Cov-2 infection in a population of negative SARS-Cov-2 hospital workers receiving preventively azithromycin, hydroxychloroquine or a Placebo

DETAILED DESCRIPTION:
Randomized clinical trial with 3 arms : hydroxychloroquine group, 300 subjects/azithromycin group, 300 subjects/ placebo of hydroxychloroquine group, 300 subjects. Hospital workers workers will be invited to participate in the study in each hospital and they will be included after giving their consent, assessment of their eligibility criteria, endonasal PCR and serolology at baseline. They will be randomized in one of the 3 arms, receive their treatment and will be followed by physical visit (at Day 2, Day 5, Day 15, Day 28) and by phone (at Day) 40 days with clinical data collection (tolerance and clinical signs of infection). At the end of treatment, another serology will be collected.

ELIGIBILITY:
Inclusion Criteria:

Hospital workers working at AP-HP hospitals over the age of 18

* Hospital workers who have signed consent
* No signs of COVID-19 infection
* Women who are likely to procreate should have a negative pregnancy test on inclusion day. In addition, they should use at least one effective contraceptive method before starting treatment, during treatment and up to 8 months after the last drug tested during the trial. Sexually active men should also have effective contraception during treatment and for at least 8 months after the last drug tested during the trial.
* Affiliated or beneficiary of Social Security

Exclusion Criteria:

* History of SARS-CoV-2 infection confirmed by PCR or serology is available at inclusion
* A history of clinical episode suspecting a PCR-confirmed or unconfirmed COVID-19 infection.
* Pregnancy and breastfeeding
* Allergy or contraindications to one of the 2 drugs in the study
* Known retinopathy
* Long congenital QT syndrome (or known in the family)
* QTc or 450 ms in men, or 460 ms in women, if Fc 55/mn (except in case of intense sport practice), if ESV on baseline ECG, if QRS - or 120 ms, if AC/FA, if the PR or BAV lengthening
* History of severe ischemic heart disease or unbalanced heart failure.
* Clinically significant bradycardia known
* Known kidney or liver failure
* Known G6PD deficit
* Subject who received antiviral treatment in the 14 days prior to inclusion
* Subject who had treatment with azithromycin or hydroxychloroquine, in the 14 days prior to inclusion
* Hypokaliemia (<= 3.5 mmol/L), Increase in creatinine (>=120 micromol/Ll, Increase in transaminases at baseline (>=2N)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
To assess the impact of hydroxychloroquine and azithromycin on the prevention of SARS-CoV-2 contamination in hospital workers exposed to 40 days of treatment. | 3 months
  The number of hospital workers with a positive serology or a positive PCR within 40 days of follow-up.

SECONDARY OUTCOMES:
Reducing clinical episodes due to suspected SARS-2 CoV infection confirmed by PCR | 40 days
  Clinical signs suggesting SARS-2 CoV infection confirmed by positive endonasal PCR
Reducing seroconversion for SARS-CoV-2 without any clinical sign | 3 months
  number of seroconversion by serology between Day 0 and Day 40.
Evaluation of drug tolerance in the study | 40 days
  number of cardiological severe adverse events assessed (ECG abnormalities : widening QT, ventricular arythmia, and cardiac arrests), other serious adverse events including hospitalizations, and deaths
Evaluation on work stopping of hospital workers | 40 days
  Number of work stoppages over the period
Observance of treatment measured by plasmatic concentrations of hydroxychloroquine or azythromycine | 40 days
  Plasmatic concentrations of treatments
Incidence of cardiologic events | 40 days
  number of cardiac events, especialy ECG abnormalities (widening QT) due to treatments

CONTACTS AND LOCATIONS:
Overall Officials: Jean Ma Treluyer, MD PhD, Principal Investigator — Assitance publique - Hôpitaux de Paris.
Locations (8):
- France (8):
  - Hopial Avicenne, Bobigny
  - Hôpital GHU Paris Saclay, Le Kremlin-Bicêtre
  - Hôpital Saint Antoine, Paris
  - Hôpital Broca, Paris
  - Hôpital La Pitié-Salpétrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital européen Georges Pompidou, Paris
  - Hôpital Necker, Paris

IPD SHARING:
Plan to Share IPD: No